CLINICAL TRIAL: NCT05119023
Title: Determining the Implicit and Rule-based Learning Ability of Individuals With Aphasia to Better Align Learning Ability and Intervention
Brief Title: Determining Learning Ability in People With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sofia Vallila Rohter, Associate Professor, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021p000033; R21DC019203 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-12 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Characterization of learning (Experimental): All participants complete behavioral (computer-based) learning tasks that measure their ability to learn observationally (observational learning ability: SRT Observational learning and AGL observational learning) and via rules (rule-based AGL learning ability, [RB AGL]). Participants additionally complete standardized cognitive-linguistic tests. Learning tasks and cognitive linguistic tests are completed over the course of 2 to 3 sessions, each lasting around 2 hours each. The AGL Observational task was always completed before the rule-based AGL task. SRT Observational and AGL Observational task order was counterbalanced.
  Enrolled participants who were safe to scan via magnetic resonance imaging (MRI) completed a structural MRI scan between one-month and five months from behavioral testing of learning.
  Interventions: Behavioral: SRT Observational Learning; Behavioral: AGL Observational Learning; Behavioral: AGL Rule-based Learning; Behavioral: Standardized cognitive-linguistic assessment; Other: Brain imaging

INTERVENTIONS:
Behavioral: SRT Observational Learning — All participants completed a computer-based serial response time (SRT) task intended to measure observational (implicit) learning ability. The SRT Observational learning task is a classic paradigm, which has been integral to the understanding of implicit learning (see Schwarb & Schumacher, 2012). The current task is a replication of classic SRT tasks first described by Nissen and Bullemer (1987), adapted for eye-tracking by Kinder et al. (2008). In this task, participants look at a dot move from one of 4 positions on a computer screen. Unbeknownst to participants, dot movement followed a 12-movement pattern for most experimental blocks. Eye-tracking data is collected and eye fixations within regions of interest trigger trial advancement. Learning ability is evaluated as a comparison of saccadic response times during sequenced trials relative to pseudorandomized trials.
Behavioral: AGL Observational Learning — All participants completed a computer-based observational artificial grammar learning (AGL) task. The AGL Observational learning task is another classic test of implicit learning involving learning of ordered items through exposure (Schuchard & Thompson, 2017). Artificial grammars contain hierarchal dependencies, similar to the rules that govern word-order and syntax in natural language. In this task, participants look at sequences of geometric shapes on a computer screen. Participants judged if two sequences matched or did not match. After training, participants are shown sequences and must judge if sequences adhere to the pattern or not.
Behavioral: AGL Rule-based Learning — All participants completed a computer-based rule-based learning task intended to measure rule-based (explicit) learning ability of an artificial grammar expressed in nonlinguistic form (sequences of shapes). In this task, participants look at sequences of geometric shapes on a computer screen. Through visuals and verbal instruction, they are taught 5 rules that govern sequences. After learning rules, participants are asked to judge via button press whether novel sequences adhere to rules or not.
Behavioral: Standardized cognitive-linguistic assessment — Participants completed standardized cognitive-linguistic assessments that evaluate their ability to produce and understand language and evaluate cognitive skills of attention, executive function and working memory important for learning. Tests involve paper and pencil, looking at pictures, listening to words, indicating responses on a keyboard and talking.
Other: Brain imaging — Enrolled participants who were safe to scan via magnetic resonance imaging (MRI) completed a structural MRI scan between one-month and five months from behavioral testing of learning.

SUMMARY:
Aphasia is an impairment in the expression or comprehension of language that results from stroke, traumatic brain injury or progressive neurological disease. Approximately two million people in the United States suffer from aphasia, which has profound impacts on quality of life, the ability to return to work and participation in life activities. Research has shown that speech-language therapy, the treatment for aphasia, can significantly improve people's ability to communicate. However, a major limitation in the field of aphasia rehabilitation is the lack of predictability in patients' response to therapy and the inability to tailor treatment to individuals. Currently, aphasia treatments are selected largely based on patient's language abilities and language deficits with little consideration of learning ability, which this study refers to as learning phenotype. Learning phenotype has been used to inform rehabilitation approaches in other domains but is not currently considered in aphasia. The overarching hypothesis of this work is that poor alignment of learning ability and language therapy limits progress for patients and presents a barrier to individualizing treatment.

The objectives of the proposed study are to (1) determine the learning phenotype of individuals with aphasia, and (2) examine how lesion characteristics (size and location of damage to the brain), language ability and cognitive ability relate to learning ability. To accomplish objectives, investigators propose to measure implicit (observational) and explicit (rule-based) learning ability in people with aphasia via computer-based tasks. Regression models will be used to examine brain and behavioral factors that relate to learning ability.

DETAILED DESCRIPTION:
Aphasia is an impairment in the expression or comprehension of language that can limit people's ability to communicate needs, reduce comprehension in complex environments, and prevent a return to work or limit participation in everyday life activities. An approximate 795,000 individuals suffer from strokes each year, with 25% to 40% resulting in aphasia. The process of aphasia rehabilitation engages many mechanisms of learning as patients are guided to relearn, reaccess or regain functional use of language via therapies that involve stimuli, tasks, cues, and feedback. Currently however, clinicians base decisions about the tasks and targets of treatment methods on language deficits, and the strength and weakness of learning systems is rarely, if ever, considered. The understanding of learning in aphasia and the way that learning influences treatment outcomes is incomplete and presents a barrier in the ability for clinicians to individually tailor treatment and reliably predict outcomes.

An in-depth characterization of learning in aphasia is important, as research has suggested that multiple learning systems exist. Furthermore, manipulations to stimuli, task, and feedback can lead to differential recruitment of learning systems and unlock learning potential, particularly in clinical populations. Prior work in aphasia supports the hypothesis that individuals with aphasia suffer from impaired learning mechanisms and are sensitive to task manipulations. Such findings demonstrate that that people with aphasia (PWA) are successful learning in some conditions and not others and provides the rationale for the proposed series of studies focused on characterizing learning abilities in individuals with aphasia.

The current project proposes to use a single-subject experimental design to determine the behavioral learning phenotype of individuals with aphasia subsequent to stroke. Implicit (observational) and explicit (rule-based) learning is quantified in individuals with aphasia using short computer-based experimental tasks. Investigators additionally explore whether effect size of learning under observational and rule-based conditions is predicted by lesion characteristics (size and extent of brain damage in regions of interest), cognitive abilities (such as attention, working memory, executive function) and language severity. Findings will help establish the behavioral and biological validity of learning phenotypes in aphasia and will provide essential information needed to support future treatment studies that align learning ability and language therapy to promote enhanced outcomes.

Overall Study Design The study will be conducted at the Massachusetts General Hospital (MGH) MGH-Institute of Health Professions. Structural scans will be obtained at the MGH Athinoula A. Martinos Biomedical Imaging Center. Participants with aphasia subsequent to stroke, in the chronic stages of their aphasia (at least 6 months post-stroke) will be recruited to participate. All participants will complete standardized assessments of cognitive and language abilities and will complete computer-based tasks evaluating observational and rule-based learning ability. Structural scans will be obtained to quantify the presence brain damage in parts of the brain that are thought to relate to learning. A key novelty of the approach is to introduce an evaluation of learning ability into diagnostic models of aphasia, incorporating subject-specific behavioral and neural metrics.

ELIGIBILITY:
Inclusion criteria

* Aphasia due to left hemisphere stroke
* Must be in the chronic stages of aphasia, at least 6 months post onset of stroke
* Must be between the ages of 18 and 80 years of age
* Must have near to normal uncorrected or corrected vision per self-report
* Must be medically and neurologically stable and at least wheelchair ambulatory

Exclusion criteria

* History of significant psychiatric or medical disease
* Presence of visual field cuts or visual neglect as determined by the Cognitive Linguistic Quick Test (CLQT; Helm-Estabrooks, 2017) symbol cancellation task
* Implanted medical devices or metal fragments that are not MRI safe

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Vallila-Rohter, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Institute of Health Professions, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets, statistical analysis codes and experimental set-ups with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with NIH policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Ashby FG, Alfonso-Reese LA, Turken AU, Waldron EM. A neuropsychological theory of multiple systems in category learning. Psychol Rev. 1998 Jul;105(3):442-81. doi: 10.1037/0033-295x.105.3.442. PMID 9697427
- [Background] Ashby FG, O'Brien JB. Category learning and multiple memory systems. Trends Cogn Sci. 2005 Feb;9(2):83-9. doi: 10.1016/j.tics.2004.12.003. PMID 15668101
- [Background] Davis T, Love BC, Maddox WT. Two pathways to stimulus encoding in category learning? Mem Cognit. 2009 Jun;37(4):394-413. doi: 10.3758/MC.37.4.394. PMID 19460948
- [Background] Shohamy D, Myers CE, Onlaor S, Gluck MA. Role of the basal ganglia in category learning: how do patients with Parkinson's disease learn? Behav Neurosci. 2004 Aug;118(4):676-86. doi: 10.1037/0735-7044.118.4.676. PMID 15301595
- [Background] Squire LR, Knowlton BJ. Learning about categories in the absence of memory. Proc Natl Acad Sci U S A. 1995 Dec 19;92(26):12470-4. doi: 10.1073/pnas.92.26.12470. PMID 8618923
- [Background] Vallila-Rohter S, Kiran S. Non-linguistic learning and aphasia: evidence from a paired associate and feedback-based task. Neuropsychologia. 2013 Jan;51(1):79-90. doi: 10.1016/j.neuropsychologia.2012.10.024. Epub 2012 Nov 2. PMID 23127795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with aphasia were recruited by referral from physicians, speech-language pathologists, neuropsychologists. Individuals with aphasia were also recruited from the MGH-Institute of Health Professions Aphasia Center. Participants were recruited via word of mouth, flyers/presentations and through Rally at Mass General Brigham, an online portal advertising research studies being carried out within the Mass General Brigham Network. The recruitment period lasted from 5/15/22 - 7/15/23
Period: Characterization of Learning-visits 1&2
Arm/Group | Characterization of Learning
Started | 18
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Change in health status unrelated to study rendered unable to participate | 2
Not completed — Lost to Follow-up | 1
Period: Brain Imaging - Session 3
Arm/Group | Characterization of Learning
Started (Eight of the consented participants who completed period 1 (characterization of learning) were MR-safe and completed a structural brain scan between one-month and five months from behavioral testing of learning.) | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Characterization of Learning: All participants are assigned to complete behavioral (computer-based) learning tasks that measure their ability to learn observationally (observational learning ability) and via rules (rule-based learning ability).
  Observational Learning: All participants will complete a computer-based serial response time task intended to measure observational (implicit) learning ability. In this task, participants look at a dot move from one of 4 positions on a computer screen. Unbeknownst to participants, dot movement followed a 12-movement pattern for most experimental blocks. Eye-tracking data is collected and eye fixations within regions of interest trigger trial advancement. Learning ability is evaluated as a comparison of saccadic response times during sequenced trials relative to pseudorandomized trials.
  Rule-based Learning: All participants will complete a computer-based rule-based learning task intended to measure rule-based (explicit) learning ability. In this task, participants look at sequences of geometric shapes on a computer screen. Through visuals and verbal instruction, they are taught 5 rules that govern sequences. After learning rules, participants are asked to judge via button press whether novel sequences adhere to rules or not.
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.89 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18
Months post stroke [Mean (Standard Deviation); unit: Months] | 106 (96.2)

OUTCOME MEASURES:

1. Primary Outcome: SRT Observational Learning Ability
Description: For the SRT observational learning task, responses are made via eye gaze into a visual area of interest (AOI). Reaction times (RTs) are recorded as the time between target onset and gaze fixation within the target AOI. A trial is considered incorrect if an eye fixation was made that does not correspond to the target AOI. RTs for correct trials are examined. Outlier RTs three standard deviations above the mean RT of each block are removed. A score of learning is computed by comparing RTs on the last (7th) sequenced block of trials with RTs on the following (8th) pseudorandomized block (Schwarb & Schumacher, 2012). A Cohen's d effect size (ES) of observational learning is calculated for each individual participant that compares mean RTs on the final sequenced block (S7) and the pseudorandom block (PS8) using pooled standard deviations. Mean Cohen's d is reported. Negative values indicate better learning.
Time Frame: Study visit 1 or 2, AGL Observational task completed before rule-based AGL task. SRT Observational and AGL Observational task order counterbalanced
Measure: Mean (Standard Deviation); unit: Cohen's d
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
Cohen's d | -0.03 (0.34)

2. Primary Outcome: AGL Observational Learning Ability
Description: For the AGL Observational learning task, a percent accuracy score is computed for the test phase. Higher scores indicate better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent accuracy
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
Percent accuracy | 50.08 (12.19)

3. Primary Outcome: AGL Rule-based Learning Ability
Description: For the rule-based AGL task, a percent accuracy score is computed for the test phase. Higher scores indicate better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent accuracy
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
Percent accuracy | 63.1 (21.6)

4. Secondary Outcome: Standardized Assessment of Cognitive Linguistic Ability - Language Severity
Description: Standardized measure of severity of expressive and receptive language deficits (Western Aphasia Battery [WAB] score range 0 - 100 with high scores indicating lower severity)
Time Frame: Study visit 1 or 2
Measure: Mean (Standard Deviation); unit: units on a scale of 100
Groups:
- Characterization of Learning: All participants are assigned to complete behavioral (computer-based) learning tasks that measure their ability to learn observationally (observational learning ability) and via rules (rule-based learning ability).
  Observational Learning: All participants will complete a computer-based serial response time task intended to measure observational (implicit) learning ability. In this task, participants look at a dot move from one of 4 positions on a computer screen. Unbeknownst to participants, dot movement followed a 12-movement pattern for most experimental blocks. Eye-tracking data is collected and eye fixations within regions of interest trigger trial advancement. Learning ability is evaluated as a comparison of saccadic response times during sequenced trials relative to pseudorandomized trials.
  Rule-based Learning: All participants will complete a computer-based rule-based learning task intended to measure rule-based (explicit) learning ability. In this task, participants look at sequences of geometric shapes on a computer screen. Through visuals and verbal instruction, they are taught 5 rules that govern sequences. After learning rules, participants are asked to judge via button press whether novel sequences adhere to rules or not.
  Participants also completed standardized assessment of cognitive linguistic ability to examine the relationship between aphasia and learning
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
units on a scale of 100 | 80.5 (13.8)
Statistical Analysis 1: Comparison: Characterization of Learning; Examination of Language Severity and Characterization of learning: SRT Observational Learning Scores; Test type: Other; p = 0.39, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Characterization of Learning; Examination of Language severity and Characterization of learning: AGL Observational Learning Scores; Test type: Other; p < 0.01, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Characterization of Learning; Examination of Language severity and Characterization of learning: AGL Rule-based Learning Scores; Test type: Other; p = 0.95, Pearson's correlation — The threshold for statistical significance was p = 0.05

5. Secondary Outcome: Standardized Assessment of Cognitive Linguistic Ability - Cognitive Composite : Attention
Description: Composite scores based on standardized assessments of attention, working memory, and executive function were computed. Each score is computed and reported as an percent score. Minimum score is 0, maximum is 100. Higher scores indicate better cognitive ability.
Time Frame: Study visit 1 or 2
Measure: Mean (Standard Deviation); unit: percent score
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
percent score | 88.77 (21.87)
Statistical Analysis 1: Comparison: Characterization of Learning; Examination of Attention and Characterization of learning: SRT Observational Learning Scores; Test type: Other — Sample underpowered for regression so correlation examined; p = 0.36, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Characterization of Learning; Examination of Attention and Characterization of learning: AGL Observational Learning Scores; Test type: Other; p = 0.09, Pearson's correlation; The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Characterization of Learning; Examination of Attention and Characterization of learning: AGL Rule Based Learning; Test type: Other; p = 0.32, Pearson's correlation — The threshold for statistical significance was p = 0.05

6. Secondary Outcome: Standardized Assessment of Cognitive Linguistic Ability - Cognitive Composite : Working Memory
Description: as for outcome 5
Time Frame: Study visit 1 or 2
Measure: Mean (Standard Deviation); unit: percent score
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
percent score | 51.06 (20.67)
Statistical Analysis 1: Comparison: Characterization of Learning; Examination of Working Memory and Characterization of learning: SRT Observational Learning Scores; Test type: Other — Sample underpowered for regression so correlation examined; p = 0.64, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Characterization of Learning; Examination of Working Memory and Characterization of learning: AGL Observational Learning Scores; Test type: Other; p = 0.01, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Characterization of Learning; Examination of Working Memory and Characterization of learning: AGL Rule-based Learning Scores; Test type: Other; p = 0.79, Pearson's correlation

7. Secondary Outcome: Standardized Assessment of Cognitive Linguistic Ability - Cognitive Composite : Executive Function
Description: as for outcome 5
Time Frame: Study visit 1 or 2
Measure: Mean (Standard Deviation); unit: percent score
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 14
percent score | 75.24 (17.11)
Statistical Analysis 1: Comparison: Characterization of Learning; Examination of Executive Function and Characterization of learning: SRT Observational Learning Scores; Test type: Other — Sample underpowered for regression so correlation examined; p = 0.90, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Characterization of Learning; Examination of Executive Function and Characterization of learning: AGL Observational Learning Scores; Test type: Other; p = 0.09, Pearson's correlation — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Characterization of Learning; Examination of Executive Function and Characterization of learning: AGL Rule-based Learning Scores; Test type: Other; p = 0.24, Pearson's correlation

8. Secondary Outcome: Percent Spared Tissue Per ROI
Description: Lesion maps, in which the lesioned voxels are assigned a binary value (1 or 0), are normalized from native to the Montreal Neurological Institute (MNI) template (a standard brain template utilized in imaging studies). Individualized lesion maps are subtracted from each brain region of interest (ROI) to yield the volume of spared tissue per ROI. The percentage of spared tissue in each region is calculated by dividing the volume of spared tissue by the total volume of the MNI template atlas ROI. Two ROIs have been selected based on prior research showing differential activation in observational versus rule-based learning: the prefrontal cortex and the striatum.
Time Frame: Study visit 3, between one-month and five months from behavioral testing of learning
Measure: Mean (Standard Deviation); unit: Percent Spared Tissue within the ROI
Arm/Group | Characterization of Learning
Number analyzed (Participants) | 8
Percent Spared Tissue within the ROI
  Prefrontal cortex ROI | 88.8 (11.8)
  Striatum ROI | 79.37 (18.84)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Risks
Arm/Group | Characterization of Learning
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Due to the COVID pandemic and institutional policies related to data collection from human subjects, particularly vulnerable populations such as those having experienced a stroke, in-person data collection was delayed for this study. As a result, the sample size is smaller than initially proposed. Due to this more limited sample size, carrying our regression analyses was not appropriate, however, data are sufficient to identify the presence of individualized learning profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05119023/Prot_SAP_001.pdf